CLINICAL TRIAL: NCT02994758
Title: Development of Diagnostics and Treatment of Urological Cancers
Acronym: DEDUCER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Antti Rannikko, Senior consultant, urology, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: None yet
Record Dates: First submitted 2016-12-01; First posted 2016-12-16 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Prostate Carcinoma; Kidney Cancer; Urothelial Carcinoma; Testicular Cancer; Penile Cancer
Keywords: Prostate; bladder; renal; NGS; DSRT; drug screening; sequencing; personalised medicine
MeSH Terms: conditions — Prostatic Neoplasms; Kidney Neoplasms; Carcinoma, Transitional Cell; Testicular Neoplasms; Penile Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalised medicine arm (Other): This is a prospective "n-of-1" type of trial where every patient is his/her own control. This is a study further developing the translational use of an existing framework and infrastructure for systematic sample collection an analytics previously established in the HUB project incorporating NGS and DSRT into clinical care.
  Interventions: Other: Personalised treatment

INTERVENTIONS:
Other: Personalised treatment — Treatment based on NGS or DSRT

SUMMARY:
The purpose of the study is to evaluate whether state-of-the-art technologies such and next generation sequencing and drug sensitivity and resistance testing of patient derived tumour tissue can facilitate research translation and improve outcome of urologic cancers.

DETAILED DESCRIPTION:
Access to high-quality clinical patient material (e.g. tissue of primary tumor and metastasis, plasma and urine) linked to comprehensive registry and clinical data and molecular characterization of the patient material using state-of-the-art technologies (e.g. NGS, transcriptomics, imaging, DSRT) will facilitate a more rapid translation of basic research innovations into clinical care (diagnostics, imaging, therapeutics) and result in improved outcome of patients suffering from urologic cancers ("personalized medicine").

The principal aim of the project is to establish a framework and infrastructure for the systematic collection and interpretation of biological patient samples. Similarly, the investigators aim to establish the format how the related clinical and research data can be made readily accessible for both clinicians and researchers without compromising patient privacy. The key objectives of the project are to facilitate research translation and to improve outcome of urologic cancers.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is able to provide written informed consent and is at least 18 years of age
2. The patient must have a verified diagnosis of an urologic cancer by a board-certified clinician

Exclusion Criteria:

1. The patient is not willing to provide a written informed consent
2. The patient has a severe psychiatric illness, imprisonment or mental impairment inflicting on ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-11-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Successful clinical translation | Up to 24 months
  The magnitude of successful clinical translation is measured by the number of times project-derived personalized medicine has impacted patients care by application of novel and existing biomarkers and therapies (e.g. sequencing, DSRT) by 2020

SECONDARY OUTCOMES:
Successful pre-clinical translation | Up to 24 months
  Successful pre-clinical translation, the magnitude of which is measured by the number of times project-derived potential druggable targets or able to re-purpose treatment options were identified within the project by 2020.
Translation of preclinical data into clinically useful data. | Up to 24 months
  Translation of preclinical data into clinically useful data. The success of which is measured by the number of times preclinical data (e.g. sequencing, DSRT) was transformed into clinically useful form within 4 weeks from the time the initial sampling of the specimen was done.
Number of representative cell models developed from clinical samples. | Up to 24 months
  Representativeness is based on the genetics of the cell model and the parental tumor

CONTACTS AND LOCATIONS:
Overall Officials: Antti S Rannikko, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Saeed K, Rahkama V, Eldfors S, Bychkov D, Mpindi JP, Yadav B, Paavolainen L, Aittokallio T, Heckman C, Wennerberg K, Peehl DM, Horvath P, Mirtti T, Rannikko A, Kallioniemi O, Ostling P, Af Hallstrom TM. Comprehensive Drug Testing of Patient-derived Conditionally Reprogrammed Cells from Castration-resistant Prostate Cancer. Eur Urol. 2017 Mar;71(3):319-327. doi: 10.1016/j.eururo.2016.04.019. Epub 2016 May 6. PMID 27160946
- [Result] Saeed K, Ojamies P, Pellinen T, Eldfors S, Turkki R, Lundin J, Jarvinen P, Nisen H, Taari K, Af Hallstrom TM, Rannikko A, Mirtti T, Kallioniemi O, Ostling P. Clonal heterogeneity influences drug responsiveness in renal cancer assessed by ex vivo drug testing of multiple patient-derived cancer cells. Int J Cancer. 2019 Mar 15;144(6):1356-1366. doi: 10.1002/ijc.31815. Epub 2018 Nov 4. PMID 30125350